#### Forespørsel om deltakelse i forskningsprosjektet:

"Studiet av potensiell normalisering av hjerterytme etter medikamentbytte fra kimerisk metadon til aktivt metadon" (kortnavn MePhaCard)

# Bakgrunn og hensikt

Dette er et spørsmål til deg om å delta i en forskningsstudie for å studere grad av redusert ledningstid i hjertet (såkalt QT-tid) ved bytte fra din nåværende metadon (eksempel Metadon DNE® eller apotekfremstilt metadon) til L-metadon produsert av DNE®. Sistnevnte preparat er registrert for bruk i substitusjonsbehandling i Tyskland under navnet Polamydon og inneholder kun den aktive formen for metadon.

Undersøkelsen er et samarbeidsprosjekt mellom Avdeling for farmakologi og Spesialiserte ruspoliklinikker ved Oslo Universitetssykehus, HF.

#### Hva innebærer studien?

Du er LAR-pasient og bruker metadon og har tidligere fått påvist forlenget ledningstid (QT-tid) i hjertet. Registrerte metadonpreparater i Norge består av to typer metadon som er speilvendte i forholdt til hverandre (såkalt rasemisk metadonløsning). Disse kalles L-metadon og D-metadon (*L-metadon kalles også R-metadon, og D-metadon kalles S-metadon*). Forenklet kan man sammenligne D- og L-metadon med høyre og venstre hånd, som passer til hver sin hanske. L-metadon er den biologisk aktive formen som binder seg til opiatreseptoren i hjernen og lindrer smerter og/eller abstinenssymptomer. Foreløbige forskningsdata tyder på at D-metadon kan øke hjertets QT-tid ved binding til egne ionekanaler i hjertet. En slik forlengelse er kjent bivirkning for flere av opiatene og kan i enkelt-tilfeller medføre hjerterytmeforstyrrelser og mulig hjertestans.

Vi ønsker å undersøke grad av normalisert QT-tid ved medikamentendring fra rasemisk metadon til L-metadon. Dersom resultatene viser at L-metadon har mindre påvirkning på hjertets QT-tid, vil du kunne fortsette med dette preparatet etter endt studie.

<u>Undersøkelser under studien:</u> Det vil det gjennomføres prøvetaking og forskningsintervjuer/kartlegginger før, under og etter medikamentbytte fra rasemisk metadon til L- metadon. Disse omhandler:

- EKG for måling av hjertets ledningstid (QT-tid),
- Blodprøver for bestemmelse av metadonkonsentrasjon i serum, bestemmelse av blodsalter som er av bedtyning for hjerterytmen og skreening for relevante arvelige markører for enzymer som forbrenner metadon i kroppen og for ionekanaler i hjertet ved lang QT-tid.
- Urinprøver som normalt, eneste forskjellen er at resultatene fra disse blir brukt i undersøkelsen. For pasienter som per i dag ikke avlegger urinprøver, vil det måtte avlegges en urinprøve per 14. dag i studieperioden. Dette for å dokumentere rusmestringsmessig stabilitet.
- Forskningsintervjuer inneholder skjema som måler eventuelle abstinenssymptomer (Clinical Opioid Withdrawal Scale) og symptomer på lang QT-tid som besvimelse/nærbesvimelse og hjertebank.

# Mulige fordeler og ulemper

Forventede fordeler med deltakelsen i studien er redusert medikamentpåvirkning av hjertet, med kortere ledningstid (QT-tid) og mindre risiko for utvikling av hjerterytmeforstyrrelse.

Ulemper kan være relatert til bivirkninger forbundet med smakstilsetnignsstoffene i L-Metadon, ubehag forbundet med blodprøvetaking, EKG-taking og spørresskjema som er ulemper knyttet til din tidsbruk.

# Hva skjer med prøvene og informasjonen om deg

Prøvene tatt av deg og informasjonen som registreres om deg skal kun brukes slik som beskrevet i hensikten med studien. Alle opplysningene og prøvene vil bli behandlet konfidensielt og hver pasient vil bli gitt en nummerkode. Koden knytter deg til dine opplysninger og prøver gjennom en navneliste.

Det er kun autorisert personell knyttet til prosjektet som har adgang til navnelisten og som kan finne tilbake til deg. Det vil ikke være mulig å identifisere deg i resultatene av studien når disse publiseres.

# Frivillig deltakelse

Det er frivillig å delta i studien. Du kan når som helst og uten å oppgi noen grunn trekke ditt samtykke til å delta i studien. Dette vil ikke få konsekvenser for din videre behandling. Dersom du ønsker å delta, undertegner du samtykkeerklæringen på siste side. Om du nå sier ja til å delta, kan du senere trekke tilbake ditt samtykke uten at det påvirker din øvrige behandling. Dersom du senere ønsker å trekke deg eller har spørsmål til studien, kan du kontakte overlege Peter Krajci tlf 99 50 10 47 eller overlege Mimi Stokke Opdal tlf 23 02 62 61 ved Oslo Universitetssykehus.

**Ytterligere informasjon om studien finnes i kapittel** *A – utdypende forklaring av hva studien innebærer.* 

Ytterligere informasjon om biobank, personvern og forsikring finnes i kapittel B – *Personvern, biobank, økonomi og forsikring.* 

Samtykkeerklæring følger etter kapittel B.

# Kapittel A- utdypende forklaring av hva studien innebærer

#### Kriterier for deltakelse

For at du skal kunne delta i studien må du oppfylle følgende kriterier:

- 1. Stabilisert på fast metadondose
- 2. Fri for bruk av andre rusmidler
- 3. Påvist forlengelse av hjertets ledningstid (QT-tid), verdi over 450 ms.
- 4. Alder 18 år eller eldre
- 5. Signere skiftlig informert samtykke

Man kan ikke delta i studien dersom man oppfyller følgende kriterier:

- 1. Dersom du ikke kan møte opp til daglige observerte inntak
- 2. Dersom du bruker stoffer eller rusmidler
- Dersom du har alvorlige psykiatriske diagnoser eller ubehandlede alvorlige somatiske sykdommer, hvor symptomene og medisinering kan komplisere tolkningen av testresultatene
- 4. Dersom du er gravid

# Bakgrunnsinformasjon om studien

Halvparten av norske ca 7000 LAR-pasienter behandles med en rasemisk blanding av L- og D-metadon. L-metadon bindes 12x sterkere enn D-metadon til opiatreseptorer og behandler abstinens. D-metadon påvirker hjertemusklenes ionekanaler i sterkere grad enn L-metadon. Effekten synes å være en doseavhengig, med forlenget ledningstid (QTc-tid). Den er videre forbundet med hjerterytmeforstyrrelser og plutselig hjertestans. Norsk studie viste forlenget QTc-tid (>450 ms) hos 28,9 % av LAR-pasientene. I alt 15 LAR pasienter skal delta i studien.

#### Vitenskapelig betydning:

Medikamentbytte fra L,D- til L-metadon kan være et verdifult bidrag i tryggere behandling av pasienter med risiko for utvikling av alvorlige rytmeforstyrrelser.

#### Undersøkelser, blodprøver og annet den inkluderte må gjennom

Følgende undersøkelser (både fysiske og spørreskjemaer) er inkludert i studien:

- Elektrokardiogram (EKG)
- Blodprøver for måling av blodsalter, konsentrasjonen av metadon og relevante arvelige markører
- Vurdering av medikamenteffekt (spørreskjema for kartlegging av abstinenssymptomer)
- Vurdering av symptomer på lang QT-tid (spørreskjema)
- Rusbruk (egenrapportert og ved urinkontroll)

# Tidsskjema – hva skjer og når skjer det?

**Dag 0: Inklusjon:** Påvist QT-tid over 450 ms og du kan etter eget ønske inkluderes i studien. Det tas blodprøver av blodsalter og serumkonsentrasjon av metadon samt EKG. Du signerer samtykke skjema for frivillig deltakelse.

Dag 7-14: Daglige overvåkede inntak av metadon på apotek eller tilsvarende.

Dag 14: Oppmøte på Oslo Universitetssykehus. Du møter medikamentfastende.

# Kontroll av D,L-metadon og EKG dagen før bytte til ren L-metadon.

Utfylling av spørreskjema for kartlegging av abstinenssymptomer, lang QT-tid symptomer, blodprøver (herunder fastende metadon) og EKG før og 3 timer etter D,L-metadon inntak.

Fra dagen etter medikamentbytte fra rasemisk metadon til L-Metadon (bytteforholdet 2:1)

Dag 14-28: Daglige overvåkede inntak av **L-metadon** på apotek eller tilsvarende

Dag 28: Oppmøte på Oslo Universitetssykehus. Møter medikamentfastende. **Kontroll ved bruk av L-metadon.** 

Utfylling av spørreskjema for kartlegging av abstinenssymptomer, lang QT-tid symptomer, blodprøver (herunder fastende metadon) og EKG før og 3 timer etter L-metadon inntak.

Dag 29-42: Daglige overvåkede inntak av L-metadon på apotek eller tilsvarende

Dag 42: Oppmøte på Oslo Universitetssykehus, møter medikamentfastende. **Kontroll etter 28 dagers bruk av L-metadon.** 

Utfylling av spørreskjema for kartlegging av abstinenssymptomer, lang QT-tid symptomer, blodprøver (herunder fastende metadon) og EKG før og 3 timer etter L-metadon inntak.

# Mulige fordeler

Forventede fordeler med deltakelsen i studien er redusert medikamentpåvirkning av hjertet, med kortere ledningstid (QT-tid) og derved mindre fare for hjerterytmeforstyrrelser.

# Mulige bivirkninger

Ulemper kan være relatert til bivirkninger forbundet med smakstilsetnignsstoffene i L-Polamydon og ubehag forbundet med blodprøvetaking.

#### Mulige ubehag/ulemper

Deltakelse i studien vil kreve utvidet tidsbruk på grunn av oppmøter forbundet med prøvetaking og forskningsintervjuer.

#### Pasientens ansvar

Pasienter som velger å delta i studien forplikter seg til å følge det opplegget som studien krever. Pasientene må møte opp til riktig sted til riktig tid.

# Kompensasjon til pasienter ved gjennomført studie

Det vil <u>ikke</u> bli gitt noe kompensasjon til studiedeltakelse. Det vil bli servert drikke og rundstykker dagen på forskningsposten.

# Øvrige opplysninger

Dersom endringer skulle oppstå i studien som kan påvirke din villighet til å delta vil du informeres om dette så snart informasjon om dette er tilgengelig. Du vil også få informasjon om mulige beslutninger som gjør at deltakelse i studien kan bli avsluttet tidligere enn planlagt.

# Kapittel B - Personvern, økonomi og forsikring

#### Personvern

Opplysninger som registreres om deg er resultatet av kliniske undersøkelser med spørsmål om fornøydhet, bivirkninger, abstinensplager, rusbruk og plager (intervju SCL-25). Urinprøvene vil bli analysert rutinemessig som for andre pasienter i LAR. Alle som får innsyn i dataene har taushetsplikt. Dette inkluderer urinprøvesvar.

Oslo universitetssykehus ved administrerende direktør er databehandlingsansvarlig.

#### Rett til innsyn og sletting av opplysninger om deg og sletting av prøver

Hvis du sier ja til å delta i studien, har du rett til å få innsyn i hvilke opplysninger som er registrert om deg. Du har videre rett til å få rettet eventuelle feil i de opplysningene vi har registrert. Dersom du trekker deg fra studien, kan du kreve å få slettet innsamlede opplysninger, med mindre opplysningene allerede er inngått i analyser eller brukt i vitenskapelige publikasjoner.

Studien er finansiert av Oslo universitetssykehus, Rusbehandling Midt-Norge og legemiddelprodusenten.

#### **Forsikring**

Det vil bli tegnet en standard forsikring.

Jeg bekrefter å ha gitt informasjon om studien

# Informasjon om utfallet av studien

Pasientene vil bli informert om resultatet av undersøkelsene når disse klargjort fot publisering.

# Samtykke til deltakelse i studien Jeg er villig til å delta i studien (Signert av prosjektdeltaker, dato) Stedfortredende samtykke når berettiget, enten i tillegg til personen selv eller istedenfor (Signert av nærstående, dato)

| Kapittel A og B |
|----------------------|
| MePhaCard 27.02.2015 |

-----

(Signert, rolle i studien, dato)